CLINICAL TRIAL: NCT00378989
Title: The Effectiveness and Cost-effectiveness of Health Advice and Occupational Health Intervention on Work Ability. Two Randomised Trials.
Brief Title: The Effectiveness of Health Advice and Occupational Health Intervention on Work Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evalua International (Other)
Collaborators: Mutual Pension Insurance Company Ilmarinen (Unknown); The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government); Sitra, the Finnish Innovation Fund (Other); Pfizer (Industry); Finnish Office for Health Technology Assessment, FinOHTA/Stakes (Unknown); University of Helsinki (Other)
Responsible Party: Principal Investigator, Simo Taimela, MD, Evalua International
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EVA2XRCT
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Signs and Symptoms
MeSH Terms: conditions — Signs and Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): A letter with personal feedback of the results of a health risk appraisal and invitation to a consultation at the occupational health services.
  Interventions: Behavioral: Consultation at the occupational health services
- Control (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Consultation at the occupational health services — Consultation at the occupational health services
  Arms: Intervention

SUMMARY:
Study hypotheses were 1) Classification of the risk of sickness absence can be made with questionnaires addressing self-rated health problems; 2) Occupational health intervention of the employees at 'High Risk´ of sickness absence is more effective than usual care in controlling sickness absence; 3) Health advice intervention of the employees at 'Increased Risk´ of sickness absence is more effective than usual care in controlling sickness absence; 4) The interventions are cost-effective use of resources from the societal perspective.

DETAILED DESCRIPTION:
The study design is a longitudinal cohort study with two embedded randomised trials. The risk of sickness absence is classified on the basis of self-administered questionnaires, on the basis of a priori defined cut-off limits. Two randomised trials are performed in the subgroups of 'High Risk´ and 'Increased Risk´ of sickness absence. The study is performed within one corporation in Finland. All employees with permanent job and age between 18 and 60 years are invited to participate.

The worker's own occupational nurses and physicians execute the occupational health program for workers at 'High Risk´ for sickness absence. The employees in the "High Risk" intervention group receive a personal feedback of their health survey results in a letter, in which they are also invited to a consultation at the OHS. The main purpose of the consultation, during which the individual findings of the health survey are available for the OHS professionals, is the construction of an action plan, and if appropriate, referral to a medical specialist, or psychologist. The employees in the 'High Risk´ control group receive care as usual.

The intervention for workers at 'Increased Risk´ for sickness absence is executed as medical counselling over the telephone. The employees in the 'Increased Risk´ intervention group receive a personal feedback of their questionnaire results in a letter, in which they were also invited to call the phone advice centre in order to receive medical advice. The employees in the 'Increased Risk´ control group receive care as usual.

Sickness absence data is obtained from the employer's records, the baseline covering the one-year period before the intervention and the follow-up covering the one-year period after the intervention. Sickness absences are obtained without medical diagnoses. The study participants also fill in a health questionnaire including, among other questions, healthcare utilization variables at the one-year follow-up.

We will carry out an intention to treat analysis. We will use analysis of covariance (ANCOVA) to analyse sickness absence outcomes at 12 months, with corresponding baseline values and risk / treatment group as covariates. Economic evaluation will be performed alongside the randomised controlled trial within the 'High Risk´ group.

ELIGIBILITY:
Inclusion Criteria:

* Permanent job
* Age 18 to 60 years

Exclusion Criteria:

* Pension granted

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 418 (Actual)
Dates: Start 2004-09; Primary Completion 2005-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Sickness absence during the 12-month follow-up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Simo P Taimela, MD, PhD, Principal Investigator — Evalua International
Locations (1):
- Evalua International Ltd. Oy, Espoo, Finland

REFERENCES:
- [Background] Taimela S, Laara E, Malmivaara A, Tiekso J, Sintonen H, Justen S, Aro T. Self-reported health problems and sickness absence in different age groups predominantly engaged in physical work. Occup Environ Med. 2007 Nov;64(11):739-46. doi: 10.1136/oem.2006.027789. Epub 2007 Feb 15. PMID 17303674
- [Result] Taimela S, Malmivaara A, Justen S, Laara E, Sintonen H, Tiekso J, Aro T. The effectiveness of two occupational health intervention programmes in reducing sickness absence among employees at risk. Two randomised controlled trials. Occup Environ Med. 2008 Apr;65(4):236-41. doi: 10.1136/oem.2007.032706. Epub 2007 Aug 6. PMID 17681994
- [Result] Taimela S, Justen S, Aronen P, Sintonen H, Laara E, Malmivaara A, Tiekso J, Aro T. An occupational health intervention programme for workers at high risk for sickness absence. Cost effectiveness analysis based on a randomised controlled trial. Occup Environ Med. 2008 Apr;65(4):242-8. doi: 10.1136/oem.2007.033167. Epub 2007 Oct 12. PMID 17933885
- [Result] Taimela S, Aronen P, Malmivaara A, Sintonen H, Tiekso J, Aro T. Effectiveness of a targeted occupational health intervention in workers with high risk of sickness absence: baseline characteristics and adherence as effect modifying factors in a randomized controlled trial. J Occup Rehabil. 2010 Mar;20(1):14-20. doi: 10.1007/s10926-009-9221-0. PMID 20012343